CLINICAL TRIAL: NCT00592670
Title: Hypoglycemia Associated Autonomic Failure in Type 1 DM, Question 6
Brief Title: Hypoglycemia Associated Autonomic Failure in Type 1 DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Steve Davis, Chairman of Medicine.University of Maryland, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: IRB#040912-HAAF-T1DM-Q6; DK69803
Record Dates: First submitted 2008-01-01; First posted 2008-01-14 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Baseline measures followed by a randomized 6 weeks treatment of Prozac.
  Interventions: Drug: Fluoxetine
- 2 (Placebo Comparator): Baseline followed by a 6 week randomized treatment of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine — 20 mg fluoxetine orally one per day for 1 week, 40 mg fluoxetine orally once per day for one week, 80 mg Fluoxetine orally for remaining 4 weeks of treatment
  Other Names: Prozac
  Arms: 1
Drug: Placebo — 20 mg placebo pill taken orally once per day for one week, 40 mg placebo pill taken orally one per day for one week, 80 mg placebo pill taken orally once per day for remaining 4 weeks.
  Arms: 2

SUMMARY:
It is unclear what effect selective serotonin reuptake inhibitors (SSRIs) have on hypoglycemia. Thus, the American Hospital Formulary Service recommends careful monitoring of blood glucose levels in all patients with diabetes initiating or discontinuing SSRIs (Katz et al., 1996). Because of the increased prevalence of depression in those with diabetes, it is critical to discover what affect the antidepressant therapy may have on counterregulatory responses to hypoglycemia. This study hypothesizes that chronic administration of SSRIs may result in a blunted counterregulatory response to hypoglycemia, thereby leaving individuals more susceptible to hypoglycemia.

DETAILED DESCRIPTION:
Because selective serotonin reuptake inhibitors are commonly prescribed to treat depression, it is vital to understand how these antidepressants affect hypoglycemia- the most feared complication in diabetes. This study's aim is to determine whether individuals who are chronically taking selective serotonin reuptake inhibitors have a reduced ability to defend against hypoglycemia compared to individuals not taking the medication, thus leaving them more susceptible to hypoglycemia. Both healthy volunteers and volunteers with type 1 diabetes mellitus will be studied. The results could potentially be important to diabetic patients, by demonstrating to physicians how to modify therapy for those taking antidepressants in order to avoid hypoglycemia.

The known effects of SSRI on the hypothalamo pituitary axis(HPA)may be important to the counterregulation of hypoglycemia. Prior research has demonstrated in healthy volunteers that antecedent increases in plasma cortisol result in significant blunting of neuroendocrine and autonomic responses to subsequent hypoglycemia. Thus, by activating the HPA axis, SSRIs could cause blunting of the counterregulatory response to hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* 16 (8 males, 8 females) healthy volunteers aged 18-45 yr
* 34 (17 males, 17 females) type 1 diabetes volunteers aged 18-45 yr
* Body mass index 21-30 kg • m-2
* Normal bedside autonomic function
* Normal results of routine blood test to screen for hepatic, renal, and hematological abnormalities
* Female volunteers of childbearing potential: negative HCG pregnancy test
* Volunteers over 40 years old: normal heart tracing recorded while resting and walking on the treadmill
* For those with type 1 diabetes: HbA1c > 7.0%
* For those with type 1 diabetes: had diabetes for 2-15 years
* For those with type 1 diabetes: no clinical evidence of diabetic tissue complications

Exclusion Criteria:

* Prior history of poor health: any current or prior disease condition that alters carbohydrate metabolism and prior cardiac events and/or evidence for cardiac disease
* Hemoglobin of less than 12 g/dl
* Abnormal results following screening tests
* Pregnancy
* Subjects with any indication of depression, anxiety, bipolar, panic, or eating disorders
* Subjects with a past medical history or family history of mania or bipolar disorders
* Subjects unable to give voluntary informed consent
* Subjects with a recent medical illness
* Subjects with known liver or kidney disease
* Subjects taking steroids
* Subjects taking beta blockers
* Subjects on anticoagulant drugs, anemic, or with known bleeding diseases

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2005-03; Primary Completion 2007-06 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Catecholamine measures | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N. Davis, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Briscoe VJ, Ertl AC, Tate DB, Davis SN. Effects of the selective serotonin reuptake inhibitor fluoxetine on counterregulatory responses to hypoglycemia in individuals with type 1 diabetes. Diabetes. 2008 Dec;57(12):3315-22. doi: 10.2337/db08-1000. Epub 2008 Oct 3. PMID 18835927